CLINICAL TRIAL: NCT00396929
Title: Local-Tax Trial: Local Intracoronary Administration of Paclitaxel After Stent Implantation for Prevention of Restenosis in Comparison With Stent Implantation Alone and With Implantation of a Paclitaxel-Eluting Stent
Brief Title: Efficiency of a New Therapy to Treat Stenosis of Coronary Vessels in Comparison With Two Already Admitted Therapies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Acrostak (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAX-001; 2005-001481-14
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Stable or Unstable Angina Pectoris; Myocardial Ischemia
Keywords: Paclitaxel; Restenosis; Stent; Intracoronary Dosis; Paclitaxel-eluting Stent
MeSH Terms: conditions — Angina, Unstable; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: local intracoronary dosis of Paclitaxel

SUMMARY:
The aim of the study is to examine the efficacy of Paclitaxel injection after a stent implantation in patients with stenosis in native coronary arteries to prevent restenosis in comparision with two admitted therapies.

DETAILED DESCRIPTION:
The aim of the study is to examine whether in patients with stable or instable Angina pectoris and/or documented myocardial ischemia in the presence of de-novo stenosis in native coronary arteries with a degree of stenosis between 50 % and 99 % an additional local administration of paclitaxel after implantation of a conventional stent is superior to the implantation of a conventional stent alone with respect to late lumen loss (LLL). In case of superiority it will be examined whether an additional local administration of paclitaxel after implantation of a conventional stent is not inferior to the implantation of a paclitaxel-eluting stent with respect to late lumen-luss. Is this the case, superiority will be tested.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 80, males or females
* stable or instable angina pectoris and or/ documented myocardial ischemia
* willingness and ability to adhere to the study conditions
* written informed consent after patient information
* De-novo stenosis of coronary artery with a degree of stenosis between 50% and 99%, that is accessible to PTCA
* Target vessels diameter of at least 2,5 mm and length of lesion below 18 mm

Exclusion Criteria:

* Acute myocardial infarction or still elevated CK/CK-MB after acute myocardial infarction
* known severe arrhythmias that necessitate a long term antiarrhythmic therapy
* pericarditis
* intracardiac thrombus
* Bacterial endocarditis
* Cardiopulmonary reanimation with cardiac massage within the last 6 months
* Thromboembolic accident within the last 6 months
* Severe peripheral arterial occlusive disease, that excludes the use of a 6 French catheter or that requires a special antithrombotic or anticoagulatory regime
* Manifest hyperthyreosis
* Neutrohile granulocytes less than 3000/mm3 and platelets below 100.000 or above 700.000/mm3
* Renal insufficiency with serum creatinine above 1,5 mg/L
* severe systemic hypertension despite antihypertensive medication
* other diseases which might lead to protocol violations or reduce life expectancy
* significant upper intestinal bleeding within the last 6 months
* life expectancy < 1 year
* poor general condition
* Premenopausal women, women who are postmenopausal less than 2 years
* known allergy or hypersensitivity to Paclitaxel, to one of the TAXOL-components, to one of the stent components, to acetylsalicylic acid, heparin, clopidogrel or contrast agent
* Concurrent participation or participation within the last 30 days prior to screening in another drug trial or a trial with a medical device
* absence of written declaration of consent
* inability, to understand sense and purpose of the study or not willing to keep the conditions of the study
* Bifurcation stenosis, ostium stenosis, main stem stenosis ot the target vessel
* visible thrombus in target vessel
* Severely curved or sclerosed target vessel
* complete closure of target vessel
* Severe impairment of left ventricular function with left ventricular ejection fraction of less than 30%
* Patients with expected indication for operative myocardial revascularisation within the next six months
* patients with contraindication for aortocoronary bypass operation,
* patients, who are principally not available for a second coronary angiography 6 months after stent implantation or who have a contraindication for a second coronary angiography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2005-08; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective is the angiographical determination of the late lumen loss in the stent and/or persistent area, 6 month after stent implantation. | week 26 +/- 14 days

SECONDARY OUTCOMES:
The angiographical determination of the binary restenosis rate, defined as diameter stenosis of at least 50 % in the stent and / or persistent area, 6 months after stent implantation. | week 26 +/- 14 days
The angiographical determination of the degree of stenosis, defined as percentage diameter stenosis in the stent and /or persistent area, 6 months after stent implantation. | week 26, +/- 14 days
Tthe angiographical determination of the minimal lumen diameter in the stent and / or persistent area, 6 months after stent implantation. | week 26, +/- 14 days
The 6 months after stent implantation determined combined endpoint of abrupt and subabrupt closure of the target vessel, target lesion revascularisation and major adverse cardiac events including myocardial infarction and death. | week 26, +/-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Herdeg, PD, Principal Investigator — Universitätsklinikum Tübingen, Medizinische Universitäts und Poliklinik III, Abteilung Kardiologie und Kreislauferkrankungen
Locations (1):
- Abteilung Kardiologie und Kreislauferkrankungen, Medizinische Universitätsklinik und Poliklinik III, Universitätsklinikum Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Herdeg C, Gohring-Frischholz K, Haase KK, Geisler T, Zurn C, Hartmann U, Wohrle J, Nusser T, Dippon J, May AE, Gawaz M. Catheter-based delivery of fluid paclitaxel for prevention of restenosis in native coronary artery lesions after stent implantation. Circ Cardiovasc Interv. 2009 Aug;2(4):294-301. doi: 10.1161/CIRCINTERVENTIONS.108.827865.108.827865. Epub 2009 Jul 22. PMID 20031731